CLINICAL TRIAL: NCT05370144
Title: Phase II Study of Neoadjuvant Chemoradiotherapy with Hypofractionated Radiotherapy in Patients with Esophageal and Gastroesophageal Junction Adenocarcinoma
Brief Title: A Study Involving Neoadjuvant Chemoradiotherapy with Hypofractionated Radiotherapy in Patients with Esophageal and Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NACEA
Record Dates: First submitted 2022-05-04; First posted 2022-05-11 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypofractionated neoadjuvant concurrent chemoradiotherapy (Experimental): Drug: Carboplatin and Taxol (paclitaxel)
  Patients will receive carboplatin (AUC 2) and paclitaxel (50 mg/m2) intravenously for 5 weeks on Days 1,8,15,22 and 29.
  Radiation: Hypofractionated radiation
  Interventions: Radiation: Hypofractionated radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — Hypofractionated radiation 23 Gy in 5 fractions with a simultaneous integrated boost of 26 Gy in 5 fractions to the gross tumor volume (GTV) given concurrently over 1 week during week 3 of chemotherapy.

SUMMARY:
An open-label, single-centre, non-randomized, Phase II trial in patients with esophageal adenocarcinoma. This study aims to show that delivering hypofractionated neoadjuvant concurrent chemoradiotherapy is is equally effective as conventionally fractionated neoadjuvant concurrent chemoradiotherapy.

DETAILED DESCRIPTION:
Patients with carcinoma of the esophagus or gastroesophageal junction who are suitable for curative intent trimodality therapy will receive carboplatin (AUC 2) and paclitaxel (50 mg/m2) intravenously weekly for 5 weeks. External beam RT in 5 fractions over 1 week will be delivered any time between week 3-5 of chemotherapy. Ideally patients should get radiotherapy during week 3 of chemotherapy but delivery during week 4-5 is permissible with documentation of the minor deviation. RT must start within 30 calendar days of signing the informed consent form. While restaging imaging is done as per institutional guidelines, ideally patients should get a PET/CT 6 weeks post chemoradiotherapy. Patient will then go for esophagectomy 6-12 weeks after the completion of chemoradiotherapy, but ideally at 6-8 weeks post chemoradiotherapy. Patients will be assessed for acute toxicity weekly during neoadjuvant therapy and then biweekly until esophagectomy. One month after surgery, patient will have a final clinical follow up with the radiation oncologist and review any post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven invasive adenocarcinoma of the esophagus or GEJ (Siewart type I-II)
2. Surgically resectable clinical stage T1N1-3 or T2-3N0-3 and no clinical evidence of metastatic spread are eligible (M0).
3. Maximum length (based on best information available, with EGD preferred) and width of the tumor as seen on CT not exceeding 8 cm and 5 cm respectively.
4. ECOG performance status ≤ 2
5. Patient able to begin radiation treatment within 30 calendar days of signing the informed consent form.
6. Age ≥ 18 and ≤ 80.
7. Adequate hematological, renal, hepatic and pulmonary function as defined by:

   1. Hemoglobin > 100 g/L
   2. Platelet count > 100x109/L
   3. Absolute neutrophil count > 1.5x109/L
   4. Total bilirubin ≤ 1.5x the upper limit of institutional normal
   5. Creatinine ≤ 120 µmol/L
   6. FEV1 ≥ 1.5 L
8. Patients capable of childbearing are using adequate contraception.
9. Written and informed consent of patient.

Exclusion Criteria:

1. Past or current history of malignancy other than entry diagnosis except for non-melanomatous skin cancer, or curatively treated carcinoma in situ of the cervix or a cured malignancy more than 5 years prior to enrollment
2. Previous chemotherapy and radiotherapy
3. New York heart Association Class III/IV and no history of active angina. Documented myocardial infarction within the 6 months preceding registration (pretreatment echocardiogram evidence of infarct only will not exclude patients). Patients with a history of significant ventricular arrhythmia requiring medication or congestive heart failure. History of 2nd or 3rd degree heart blocks
4. Pre-existing motor or sensory neurotoxicity greater than WHO grade 1
5. Active infection or other serious underlying medical condition which would impair the ability of the patient to receive the planned treatment
6. Dementia or altered mental status that would prohibit the understanding and giving of informed consent
7. Weight loss > 20% within 3 months of the date of screening
8. Esophageal stent
9. Pregnant or lactating patients; women of childbearing potential must have a negative serum pregnancy test within 7 days of Treatment Visit 1. Women or men of childbearing potential must use effective contraception (defined by the use of two birth control methods, which can be either two barrier methods or a barrier method plus a hormonal method to prevent pregnancy). Subjects must start using birth control from the time they have signed the Informed Consent Form prior to start of therapy until 120 days post completion of study therapy or study discontinuation, which must be documented in the eCRF.
10. Patients unfit for any treatment component, including absolute contraindications for radiotherapy or Connective Tissue Disease.
11. Unable to complete surveys in English without aid of interpreter.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2027-02-03 (Estimated); Study Completion 2028-02-03 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of delivering 5-fraction hypofractionated chemoradiotherapy | up to the Post-operative visit (60-90 days after surgery)
  Tumor regression grades and pathological complete response rates determined after one week of surgery

SECONDARY OUTCOMES:
To determine the rates of acute toxicities | up to the Post-operative visit (60-90 days after surgery)
  Safety will be determined by recording adverse events as per the CTCAE classification and grading system
To compare pathological response rates to changes in tumor FDG-PET uptake | At the time of the re-staging scan (6 weeks post chemoradiotherapy).
  Changes in tumor FDG-PET standard uptake value and total lesion glycolysis
To compare pathological response rates to changes in tumor dimensions | At the time of the re-staging scan (6 weeks post chemoradiotherapy).
  Changes in tumor dimensions on CT
To compare pathological response rates to dysphagia scores | up to the Post-operative visit (60-90 days after surgery)
  Change in dysphagia score, measured at Screening/Baseline and at the Post-operative clinical follow-up
Correlate pre- and post-chemoradiation immune microenvironment composition with the above outcome variables (pathological response, dysphagia scores, changes in FDG-PET uptake and/or tumor dimensions on CT) | At the time of the re-staging scan (6 weeks post chemoradiotherapy).
  Translational correlation between immune infiltration of biopsy and resection specimens with pathological (regression grades and response rates), clinical (dysphagia scores) and imaging (FDG-PET uptake and/or tumor dimensions on CT) outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Tom Baker Cancer Centre/Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No